CLINICAL TRIAL: NCT00482300
Title: Systematic Pelvic Lymphadenectomy Versus no Lymphadenectomy in Clinical Stage I-II Endometrial Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTC-CBM-15
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2007-06-05 (Estimated); Status verified 2007-03

CONDITIONS: Endometrial Cancer
Keywords: Histologically proved endometrial carcinoma preoperatively supposed stage I-II
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Systematic pelvic lymphadenectomy

SUMMARY:
The purpose of this trial is to determine whether the addition of systematic pelvic lymphadenectomy to hysterectomy with bilateral adnexectomy improves disease-free survival (DFS) and overall survival (OS) in patients with preoperatively supposed Stage I-II endometrial cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven endometrioid or adenosquamous endometrial carcinoma.
* Patients having myometrial invasion
* Age =/< 75 years
* Informed consent.

Exclusion Criteria:

* Serous papillary and clear cell tumors.
* Karnofsky index < 80 or severe diseases contraindicating surgery
* Concomitant neoplasia (basalioma cutis excluded)
* Distant metastasis or abdominal metastasis detected intraoperatively.
* Absence of myometrial invasion at frozen section.

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Pierluigi Benedetti Panici, Full Professor, Study Chair — Department of Obstetrics and Gynecology University La Sapienza of Rome

REFERENCES:
- [Derived] Benedetti Panici P, Basile S, Maneschi F, Alberto Lissoni A, Signorelli M, Scambia G, Angioli R, Tateo S, Mangili G, Katsaros D, Garozzo G, Campagnutta E, Donadello N, Greggi S, Melpignano M, Raspagliesi F, Ragni N, Cormio G, Grassi R, Franchi M, Giannarelli D, Fossati R, Torri V, Amoroso M, Croce C, Mangioni C. Systematic pelvic lymphadenectomy vs. no lymphadenectomy in early-stage endometrial carcinoma: randomized clinical trial. J Natl Cancer Inst. 2008 Dec 3;100(23):1707-16. doi: 10.1093/jnci/djn397. Epub 2008 Nov 25. PMID 19033573